CLINICAL TRIAL: NCT06747884
Title: Trial Readiness and Endpoint Assessment in Pediatric Myotonic Dystrophy Extension
Acronym: TREAT-EXT
Status: Recruiting | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); SUNY Research Foundation (Other); University of Minnesota (Other); Roseman University of Health Sciences (Other); University of California, San Diego (Other); University of Glasgow (Other); University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: TREAT-01-002; R01NS104010-07A1 (NIH)
Record Dates: First submitted 2024-12-13; First posted 2024-12-24 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Congenital Myotonic Dystrophy; Childhood Myotonic Dystrophy; Myotonic Dystrophy
Keywords: DM1; Childhood Myotonic Dystrophy; Congenital Myotonic Dystrophy; Myotonic Dystrophy; Myotonia; Dystrophy Myotonic; DMCRN; TREAT-EXT; TREAT CDM
MeSH Terms: conditions — Myotonic Dystrophy; Myotonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sampling will occur at baseline, month 12, and month 24 to collect DNA and RNA specimens.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Congenital myotonic dystrophy (CDM): Children with congenital myotonic dystrophy. No intervention will be administered to either group.
- Childhood Myotonic Dystrophy: Children with childhood myotonic dystrophy. No intervention will be administered to either group.

SUMMARY:
This is a natural history study to improve the types of assessments and biological samples that will be used in clinical drug trials in both congenital myotonic dystrophy and childhood myotonic dystrophy.

DETAILED DESCRIPTION:
Congenital Myotonic Dystrophy (CDM) is a multi-systemic, dominantly inherited disorder caused by a trinucleotide repeat expansion (CTGn) in the DMPK gene. Children with CDM present at birth with respiratory insufficiency, talipes equiovarus, feeding difficulties and hypotonia. There is a 30% mortality rate in the first year of life. As children grow, they are at risk for intellectual impairment, autistic features, gastrointestinal symptoms, and motor delay. Childhood onset myotonic dystrophy (ChDM) is similarly multisystem and is classified as onset after birth but before 10 years of age. It likely represents a less severe form of CDM.

Currently, there is an ongoing therapeutic trial in adults with DM1 using an antisense oligonucleotide to target the destruction of the CTG repeat. The ability to conduct this trial in children is directly limited by the lack of available data regarding appropriate clinical endpoints and biomarkers. Although the underlying mechanism is the same in adult DM1 and CDM, there are specific challenges to directly transferring outcome measures into the CDM population. First, our cross-sectional data demonstrates age-related improvement in several functional outcome measures, such as the 6-minute walk. Second, in the adult DM1 clinical trial, RNA splicing changes in the tibialis anterior muscle are a primary endpoint because they correlate with functional measures. However, our pilot data with described splicing changes does not clearly correlate with the adult clinical phenotype.

This study is designed to establish valid and reliable clinical outcome assessments for children with congenital and childhood myotonic dystrophy, and to develop biomarkers for the condition.

This study will enroll up to 200 children with CDM and ChDM at participating sites. No treatment will be administered as part of this study. Patients will receive standard of care as determined by their treating physician. Study visits will occur at Baseline, Month 12, and Month 24.

ELIGIBILITY:
Inclusion Criteria (Congenital Myotonic Dystrophy Group):

* Age 5-17 years, 11 months at enrollment. Lower age limit not applicable for participants who have completed ASPIRE-DM1 protocol. Upper age limit not applicable for participants who previously participated in TREAT-01-001 (TREAT-CDM) study
* A diagnosis of CDM, defined as: children having symptoms of myotonic dystrophy in the newborn period (<30 days), such as hypotonia, feeding or respiratory difficulty, requiring hospitalization to a ward or to the neonatal intensive care unit for more than 72 hours; and a genetic test confirming an expanded trinucleotide (CTG) repeat in the DMPK gene in the child or mother. An expanded CTG repeat size in the child is considered greater than 200 repeats or E1-E4 classification (E1= 200-500, E2=500-1,000, E3=1,000-1,500, E4>1,500).
* Written, voluntary informed consent must be obtained before any study related procedures are conducted.

Inclusion Criteria (Childhood Myotonic Dystrophy Group):

* Age 3-17 years, 11 months at enrollment. Upper age limit not applicable for participants who previously participated in TREAT-01-001 (TREAT-CDM) study.
* A diagnosis of ChDM, defined as: children having cognitive deficits, muscle weakness, myotonia that developed after age 1 and prior to age 10 and a genetic test confirming an expanded trinucleotide (CTG) repeat in the DMPK gene in the child or mother. An expanded CTG repeat size in the child is considered greater than 200 repeats or E1-E4 classification (E1= 200-500, E2=500-1,000, E3=1,000-1,500, E4>1,500).
* Written, voluntary informed consent must be obtained before any study related procedures are conducted.

Exclusion Criteria:

* Any other non-DM1 illness that would interfere with the ability to undergo safe testing or would affect the interpretation of the results, in the opinion of the site investigator
* Significant trauma within the past month
* Internal metal or devices (exclusion for DEXA component)
* Use of anticoagulants, such as warfarin or a direct oral anticoagulant (e.g., dabigatran) due to the increased risk of bleeding with biopsy
* Platelet count <50,000
* History of a bleeding disorder
* Participation in a clinical trial involving an investigational product
* History of adverse reaction to lidocaine (if participating in muscle biopsy)

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study will enroll up to 200 children with CDM and ChDM.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-06-06 (Actual); Primary Completion 2030-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Change in ambulation over 24 months as measured by the 10-Meter Walk/Run Test (10M WRT) | Baseline, Month 12 and Month 24 visits
  The participant will be timed walking or running along a 10-meter course. It is scored by recording the total time taken to ambulate 6 meters (m) is recorded to the nearest hundredth of a second. 6 m is then divided by the total time (in seconds) taken to ambulate and recorded in m/s.
Change in mobility (100-meter timed test) | Baseline, Month 12 and Month 24 visits
  Mobility will be measured using the 100 Meter Timed Test (100m) in which the participant is asked to complete 2 laps around 2 cones set 25 meters apart as quickly as safely possible, running if able. The total time in seconds is recorded from when the participant starts walking until they break the plane of the 100 meter mark (i.e., when any part of the body passes the 100 meter mark).
Change in Time to Stand (SUPINE TO STAND test) | Baseline, Month 12 and Month 24 visits
  Participant will be timed transitioning from a supine position to standing. The participant will complete one trial of this test. The test measures the participant's ability to quickly rise from a supine position on the floor with arms at their sides, to full upright posture with arms at their sides. This should be performed without external support from another person, a device, or furniture. Results will be reported in seconds.
Change in Gross Motor Function (GMFM-88) | Baseline, Month 12 and Month 24 visits
  The Gross Motor Function Measure (GMFM-88) is an assessment tool originally designed and evaluated to measure changes in gross motor function over time or with intervention in children with cerebral palsy. The GMFM assesses functional abilities including; lying/rolling, sitting, crawling/kneeling, standing, and walking/running/jumping. A four-point ordinal scale of measurement is used to assess each item, higher scores denote better performance. A score of 4 on an item indicates a consistently normal response, a score > 4 indicates persistent hypertonus, and a score < 4 indicates various degrees of hypotonus.
Change in Handheld Dynamometry and Grip HAND-HELD DYNAMOMETRY (HHD) | Baseline, Month 12 and Month 24 visits
  Maximum hand and grip strength will be assessed using a myometer. The participant will be asked to squeeze a handheld tool. When performing a hand-held dynamometry (HHD) test, you generally want a high score as it indicates greater muscle strength in the tested area; a higher number signifies a stronger muscle contraction.
9-HOLE PEGBOARD TEST (9HPT) | Baseline, Month 12 and Month 24 visits
  The Nine-Hole Peg Test (9-HPT) is a standardized, quantitative assessment used to measure finger dexterity. Test is measured in seconds.
VIDEO HAND OPENING TIME (vHOT) | Baseline, Month 12 and Month 24 visits
  . The participant will squeeze the hand for three seconds then open the hand as quickly as possible. A video recording of the procedure will be obtained showing the forearm and hand but not the face. Recordings will later be assessed by a blinded reviewer to determine the hand opening time. The time is recorded in seconds.
IOWA PERFORMANCE INSTRUMENT (IOPI) | Baseline, Month 12 and Month 24 visits
  The IOPI consists of a pressure bulb attached to a manometer. The pressure bulb will be placed on the participant's tongue. Participants are asked to push the bulb against the hard palate on the alveolar ridge just behind the upper central incisors for 3-5 seconds. This test should be repeated 3 times with a 30-second interval between trials. The maximum pressure is recorded.
CLINICAL EVALUATION OF LANGUAGE FUNDAMENTALS, 5th edition (CELF-5) | Baseline, Month 12 and Month 24 visits
  The mean score is 100, with a standard deviation of 15, meaning that standard scores between 85-115 are within the normal range. You can calculate the level of severity for delayed skills according to how many deviations below the mean a client's score is: Mild: 70-85, Moderate 55-70 , Severe: 55 and lower.
TIMED WATER SWALLOW TEST (TWST) | Baseline, Month 12 and Month 24 visits
  Participants will be given 3 ounces (90 mL) of water to drink from a clear cup. Safety of completing this test will be determined by the site PI with input from the parents/caregivers. Participants will be asked to drink the water as they normally would, without interruption. Straws may be used, if that is preferred. Participants will be asked to say aloud "I'm done" when they feel they've completed the task with a written cue provided as a reminder.26,27 Testing will be recorded for later quantification of time needed for test, volume ingested, volume/swallow, time/swallow, and swallow capacity (mL/swallow).
DOMAIN DELTA QUESTIONNAIRE | Baseline, Month 12 and Month 24 visits
  A "domain delta questionnaire" is a patient-reported questionnaire used in clinical research to assess how much a patient perceives their health status has changed across specific domains (like mobility, overall health, or upper limb function) between two points in time, essentially asking them if they feel they have gotten better, worse, or stayed the same in each area compared to a baseline measurement; it's a way to measure perceived change in health related quality of life over time.
INTELLIGIBILITY IN CONTEXT SCALE (ICS) | Baseline, Month 12 and Month 24 visits
  The ICS is a brief, 7-question, caregiver proxy instrument that rates relative intelligibility of a child with a variety of familiar and unfamiliar communication partners. It uses a 5-point Likert scale to rate the approximate level of intelligibility. ICS scores indicate a child's level of functional intelligibility, ranging from a score of 1.00 (low intelligibility) to a score of 5.00 (high intelligibility). If a child achieves an average score of 3.5, then it may be appropriate to indicate that the child is usually to sometimes understood.
PEDIATRIC QUALITY OF LIFE (PEDS QL) - GENERIC CORE SCALES | Baseline, Month 12 and Month 24 visits
  The PedsQL evaluates a child's health-related quality of life (HRQoL) with respect to social, emotional, physical, and school functioning. he PedsQL 4.0 Generic Core Scales consist of four scales measuring HRQoL in four domains: Physical, Emotional, Social, and School functioning. Scores of 81 or higher on the PedsQL™ SCD pain scales should be considered good HRQL functioning. These children likely have had less pain that was less severe than children with lower scores and/or are managing their symptoms well.
PEDIATRIC DAYTIME SLEEPINESS SCALE (PDSS) | Baseline, Month 12 and Month 24 visits
  SS is an 8-item scale that assesses daytime sleepiness in children as a PRO that has been used in sleep disordered breathing and epilepsy studies. 5 points Likert scale (0-4) for 8 questions concerning to sleepiness. Higher scores on PDSS were associated with reduced total sleep time, poorer school achievement, poorer anger control, and frequent illness.
BEHAVIOR RATING INVENTORY OF EXECUTIVE FUNCTION -2 (BRIEF2) | Baseline, Month 12 and Month 24 visits
  The BRIEF2 gives you the information you need to help children and adolescents with executive dysfunction. It digs deeper than similar measures and pinpoints exactly where and why children struggle, so therapists and schools can make informed and impactful intervention and accommodation recommendations. For all BRIEF2 clinical scales and indexes, T scores from 60 to 64 are considered mildly elevated, and T scores from 65 to 69 are considered potentially clinically elevated. T scores at or above 70 are considered clinically elevated.
VINELAND ADAPTIVE BEHAVIOR SCALES THIRD EDITION (VINELAND-3) | Baseline, Month 12 and Month 24 visits
  Vineland Adaptive Behavior Scales 3rd Edition is a leading instrument for diagnosing intellectual and developmental disabilities, providing valuable information for educational and treatment plans. Higher Internalizing and Externalizing v-scale scores indicate more problem behavior. If qualitative descriptors are desired, scores of 1 to 17 may be considered Average, 18 to 20 Elevated, and 21 to 24 Clinically Significant.
WECHSLER INTELLIGENCE SCALE FOR CHILDREN (WISC-V) | Baseline, Month 12 and Month 24 visits
  Wechsler Intelligence Scale for Children (WISC-V) is an intelligence test that measures a child's intellectual ability and 5 cognitive domains that impact performance. Low Average: 80-89. Students who test in this range may struggle to keep up in school, but are not generally eligible for special education or assistance. Average: 90-109. Students who test in this range are average and may or may not struggle to keep up in school.
AUTISM SPECTRUM SCREENING QUESTIONNAIRE (ASSQ) | Baseline, Month 12 and Month 24 visits
  Results consist of a total score between 0 and 54, where higher scores indicate that many characteristics of ASD were reported. A score of 13 and above indicates ASD is probable, with a true positive rate of 90% and a false positive rate of 22%.
REPETITIVE BEHAVIOR SCALE - REVISED (RBS-R) | Baseline, Month 12 and Month 24 visits
  The RBS-R is a questionnaire that focuses exclusively on RRBs. It includes 43 items rated on a four-point Likert scale: 0=behavior does not occur; 1=behavior occurs and is a mild problem; 2=behavior occurs and is a moderate problem; and 3=behavior occurs and is a severe problem.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Johnson, MD, MSCI, FAAN, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
Aggregated and deidentified data will be shared with qualified investigators upon majority approval of the DMCRN investigators.

REFERENCES:
- [Background] Bodfish JW, Symons FJ, Parker DE, Lewis MH. Varieties of repetitive behavior in autism: comparisons to mental retardation. J Autism Dev Disord. 2000 Jun;30(3):237-43. doi: 10.1023/a:1005596502855. PMID 11055459
- [Background] Ehlers S, Gillberg C, Wing L. A screening questionnaire for Asperger syndrome and other high-functioning autism spectrum disorders in school age children. J Autism Dev Disord. 1999 Apr;29(2):129-41. doi: 10.1023/a:1023040610384. PMID 10382133
- [Background] Huckabee ML, McIntosh T, Fuller L, Curry M, Thomas P, Walshe M, McCague E, Battel I, Nogueira D, Frank U, van den Engel-Hoek L, Sella-Weiss O. The Test of Masticating and Swallowing Solids (TOMASS): reliability, validity and international normative data. Int J Lang Commun Disord. 2018 Jan;53(1):144-156. doi: 10.1111/1460-6984.12332. Epub 2017 Jul 5. PMID 28677236
- [Background] Porter K, Smart S, Hennessey N, Cocks N. Chewing skills in two and three year old children: Gender and age comparisons on an adapted version of the test of mastication and swallowing (TOMASS-C). Int J Speech Lang Pathol. 2024 Feb;26(1):38-44. doi: 10.1080/17549507.2022.2152867. Epub 2022 Dec 13. PMID 36511843
- [Background] Frank U, van den Engel-Hoek L, Nogueira D, Schindler A, Adams S, Curry M, Huckabee ML. International standardisation of the test of masticating and swallowing solids in children. J Oral Rehabil. 2019 Feb;46(2):161-169. doi: 10.1111/joor.12728. Epub 2018 Oct 27. PMID 30307651
- [Background] Patel R, Connaghan K, Franco D, Edsall E, Forgit D, Olsen L, Ramage L, Tyler E, Russell S. "The caterpillar": a novel reading passage for assessment of motor speech disorders. Am J Speech Lang Pathol. 2013 Feb;22(1):1-9. doi: 10.1044/1058-0360(2012/11-0134). Epub 2012 Jul 30. PMID 22846881
- [Background] Berggren KN, Hung M, Dixon MM, Bounsanga J, Crockett B, Foye MD, Gu Y, Campbell C, Butterfield RJ, Johnson NE. Orofacial strength, dysarthria, and dysphagia in congenital myotonic dystrophy. Muscle Nerve. 2018 Sep;58(3):413-417. doi: 10.1002/mus.26176. PMID 29901230
- [Background] Gavazzi F, Adang L, Waldman A, Jan AK, Liu G, Lorch SA, DeMauro SB, Shults J, Pierce SR, Ballance E, Kornafel T, Harrington A, Glanzman AM, Vanderver A. Reliability of the Telemedicine Application of the Gross Motor Function Measure-88 in Patients With Leukodystrophy. Pediatr Neurol. 2021 Dec;125:34-39. doi: 10.1016/j.pediatrneurol.2021.09.012. Epub 2021 Sep 24. PMID 34624609
- [Background] McDonald CM, Marden JR, Shieh PB, Wong BL, Lane H, Zhang A, Nguyen H, Frean M, Trifillis P, Koladicz K, Signorovitch J. Disease progression rates in ambulatory Duchenne muscular dystrophy by steroid type, patient age and functional status. J Comp Eff Res. 2023 Apr;12(4):e220190. doi: 10.57264/cer-2022-0190. Epub 2023 Feb 7. PMID 36749302
- [Background] Eriksson BM, Ekstrom AB, Peny-Dahlstrand M. Daily activity performance in congenital and childhood forms of myotonic dystrophy type 1: a population-based study. Dev Med Child Neurol. 2020 Jun;62(6):723-728. doi: 10.1111/dmcn.14395. Epub 2019 Nov 8. PMID 31701525
- [Background] Johnson NE, Ekstrom AB, Campbell C, Hung M, Adams HR, Chen W, Luebbe E, Hilbert J, Moxley RT 3rd, Heatwole CR. Parent-reported multi-national study of the impact of congenital and childhood onset myotonic dystrophy. Dev Med Child Neurol. 2016 Jul;58(7):698-705. doi: 10.1111/dmcn.12948. Epub 2015 Oct 28. PMID 26510705
- [Background] Johnson NE, Butterfield R, Berggren K, Hung M, Chen W, DiBella D, Dixon M, Hayes H, Pucillo E, Bounsanga J, Heatwole C, Campbell C. Disease burden and functional outcomes in congenital myotonic dystrophy: A cross-sectional study. Neurology. 2016 Jul 12;87(2):160-7. doi: 10.1212/WNL.0000000000002845. Epub 2016 Jun 15. PMID 27306634
- [Background] Timchenko L. Correction of RNA-Binding Protein CUGBP1 and GSK3beta Signaling as Therapeutic Approach for Congenital and Adult Myotonic Dystrophy Type 1. Int J Mol Sci. 2019 Dec 21;21(1):94. doi: 10.3390/ijms21010094. PMID 31877772
- [Background] Charlet-B N, Savkur RS, Singh G, Philips AV, Grice EA, Cooper TA. Loss of the muscle-specific chloride channel in type 1 myotonic dystrophy due to misregulated alternative splicing. Mol Cell. 2002 Jul;10(1):45-53. doi: 10.1016/s1097-2765(02)00572-5. PMID 12150906
- [Background] Wagner SD, Struck AJ, Gupta R, Farnsworth DR, Mahady AE, Eichinger K, Thornton CA, Wang ET, Berglund JA. Dose-Dependent Regulation of Alternative Splicing by MBNL Proteins Reveals Biomarkers for Myotonic Dystrophy. PLoS Genet. 2016 Sep 28;12(9):e1006316. doi: 10.1371/journal.pgen.1006316. eCollection 2016 Sep. PMID 27681373
- [Background] Osborne RJ, Lin X, Welle S, Sobczak K, O'Rourke JR, Swanson MS, Thornton CA. Transcriptional and post-transcriptional impact of toxic RNA in myotonic dystrophy. Hum Mol Genet. 2009 Apr 15;18(8):1471-81. doi: 10.1093/hmg/ddp058. Epub 2009 Feb 17. PMID 19223393
- [Background] Wheeler TM. Myotonic dystrophy: therapeutic strategies for the future. Neurotherapeutics. 2008 Oct;5(4):592-600. doi: 10.1016/j.nurt.2008.08.001. PMID 19019311
- [Background] Mankodi A, Teng-Umnuay P, Krym M, Henderson D, Swanson M, Thornton CA. Ribonuclear inclusions in skeletal muscle in myotonic dystrophy types 1 and 2. Ann Neurol. 2003 Dec;54(6):760-8. doi: 10.1002/ana.10763. PMID 14681885
- [Background] Mankodi A, Takahashi MP, Jiang H, Beck CL, Bowers WJ, Moxley RT, Cannon SC, Thornton CA. Expanded CUG repeats trigger aberrant splicing of ClC-1 chloride channel pre-mRNA and hyperexcitability of skeletal muscle in myotonic dystrophy. Mol Cell. 2002 Jul;10(1):35-44. doi: 10.1016/s1097-2765(02)00563-4. PMID 12150905
- [Background] Campbell C, Sherlock R, Jacob P, Blayney M. Congenital myotonic dystrophy: assisted ventilation duration and outcome. Pediatrics. 2004 Apr;113(4):811-6. doi: 10.1542/peds.113.4.811. PMID 15060232
- [Background] Johnson NE, Luebbe E, Eastwood E, Chin N, Moxley RT 3rd, Heatwole CR. The impact of congenital and childhood myotonic dystrophy on quality of life: a qualitative study of associated symptoms. J Child Neurol. 2014 Jul;29(7):983-6. doi: 10.1177/0883073813484804. Epub 2013 Apr 22. PMID 23611887
- [Background] Campbell C, Levin S, Siu VM, Venance S, Jacob P. Congenital myotonic dystrophy: Canadian population-based surveillance study. J Pediatr. 2013 Jul;163(1):120-5.e1-3. doi: 10.1016/j.jpeds.2012.12.070. Epub 2013 Feb 14. PMID 23415617
- [Background] Johnson NE, Butterfield RJ, Mayne K, Newcomb T, Imburgia C, Dunn D, Duval B, Feldkamp ML, Weiss RB. Population-Based Prevalence of Myotonic Dystrophy Type 1 Using Genetic Analysis of Statewide Blood Screening Program. Neurology. 2021 Feb 16;96(7):e1045-e1053. doi: 10.1212/WNL.0000000000011425. Epub 2021 Jan 20. PMID 33472919
- [Background] Mahadevan M, Tsilfidis C, Sabourin L, Shutler G, Amemiya C, Jansen G, Neville C, Narang M, Barcelo J, O'Hoy K, et al. Myotonic dystrophy mutation: an unstable CTG repeat in the 3' untranslated region of the gene. Science. 1992 Mar 6;255(5049):1253-5. doi: 10.1126/science.1546325.
- [Background] Brook JD, McCurrach ME, Harley HG, Buckler AJ, Church D, Aburatani H, Hunter K, Stanton VP, Thirion JP, Hudson T, et al. Molecular basis of myotonic dystrophy: expansion of a trinucleotide (CTG) repeat at the 3' end of a transcript encoding a protein kinase family member. Cell. 1992 Feb 21;68(4):799-808. doi: 10.1016/0092-8674(92)90154-5. PMID 1310900
- [Background] Fu YH, Pizzuti A, Fenwick RG Jr, King J, Rajnarayan S, Dunne PW, Dubel J, Nasser GA, Ashizawa T, de Jong P, et al. An unstable triplet repeat in a gene related to myotonic muscular dystrophy. Science. 1992 Mar 6;255(5049):1256-8. doi: 10.1126/science.1546326.